CLINICAL TRIAL: NCT00051168
Title: A Long-term Safety Study of Once-daily TRAVATAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-02-20
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2010-04

CONDITIONS: Glaucoma, Open-angle; Ocular Hypertension
Keywords: Glaucoma; POAG; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Travoprost

ARMS (1):
- Travatan (Experimental): Travoprost (0.004%)
  Interventions: Drug: Travatan

INTERVENTIONS:
Drug: Travatan — Travoprost (0.004%) 1 drop each eye once daily

SUMMARY:
Long term safety study of TRAVATAN in patients with Open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Adult patients of any race and either sex with chronic angle-closure glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Europe, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in ophthalmic clinics, academic and civil hospitals from September 24, 2002. Last patient completed the study on March 23, 2009.
Period: Overall Study
Arm/Group | Travatan
Started | 502
Completed | 367
Not Completed | 135

BASELINE CHARACTERISTICS:
Arm/Group | Travatan
Number analyzed (Participants) | 502
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 237
  >=65 years | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281
  Male | 221

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure
Description: Mean IOP for the patient's worse eye at baseline was used in the secondary endpoint analysis. 2 consecutive IOP measurements for each eye were taken. If the 2 measurements for the same eye differ by 4 mmHg or less, the average of the measurements would be considered as the mean IOP for that eye. If the 2 measurements for the same eye differ by more than 4 mmHg, then a third measurement was to be taken.
  All IOP measurements were performed with a Goldmann applanation tonometer.
Time Frame: At 5 years.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mm Hg)
Arm/Group | Travatan
Number analyzed (Participants) | 502
millimeters mercury (mm Hg) | 16.5 (2.6)

ADVERSE EVENTS:
Time Frame: Baseline to 5 years.
Description: Adverse events were both volunteered and solicited.
Arm/Group | Travatan
Serious Adverse Events (participants affected / at risk) | 99/502
Other Adverse Events (participants affected / at risk) | 304/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travatan (N=502)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Renal failure (Renal and urinary disorders) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (5)
Cholecystectomy (Surgical and medical procedures) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Choroidal Neovascularisation (Eye disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Hip surgery (Surgical and medical procedures) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypopharyngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 8 (8)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Knee operation (Surgical and medical procedures) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung operation (Surgical and medical procedures) | 1 (1)
Lymphadenectomy (Surgical and medical procedures) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Trabeculoplasty (Surgical and medical procedures) | 1 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travatan (N=502)
Cataract (Eye disorders) | 147 (195)
Iris hyperpigmentation (Eye disorders) | 148 (151)
Hypertension (Vascular disorders) | 83 (97)
Visual acuity reduced (Eye disorders) | 55 (73)
Ocular hyperemia (Eye disorders) | 50 (56)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 38 (41)
Injury (Injury, poisoning and procedural complications) | 25 (26)
Dry eye (Eye disorders) | 25 (28)
Diabetes mellitus (Metabolism and nutrition disorders) | 26 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less